CLINICAL TRIAL: NCT04190602
Title: The AcChord Study: A Multicenter Post-Market Observational Registry of the NeoChord Artificial Chordae Delivery System
Brief Title: Multicenter Post-Market Observational Registry of the NeoChord Artificial Chordae Delivery System
Acronym: AcChord
Status: Recruiting | Type: Observational
Sponsor: NeoChord (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-610414-101
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Mitral Regurgitation; Mitral Valve Disease; Mitral Valve Insufficiency; Mitral Valve Prolapse; Heart Valve Diseases
Keywords: NeoChord; DS1000; Artificial Chordae; Mitral Valve Repair
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NeoChord Artificial Chordae Delivery System, Model DS1000 — The intended use of the device is for the placement of artificial chordae when the natural chordae tendinae have become elongated or ruptured due to degenerative valve disease.
  Other Names: NeoChord DS1000; DS1000

SUMMARY:
The objective of this study is to evaluate the 5-year outcomes of participants with degenerative mitral valve disease treated with the NeoChord Artificial Chordae System, Model DS1000 in a post-market setting.

DETAILED DESCRIPTION:
This study is an observational, single-arm, multicenter post-market registry. Both prospective and retrospective enrollment will be allowed. No additional invasive or burdensome examinations outside those routinely required for the standard mitral valve repair procedure will be requested.

ELIGIBILITY:
Inclusion Criteria:

* Has Grade III Moderate or Grade IV Severe degenerative or mixed disease mitral valve regurgitation
* Study procedure completed after 31 December 2016

Exclusion Criteria:

* Heavily calcified valves
* Valvular retraction with severely reduced mobility
* Active bacterial endocarditis
* Complex mechanism of MR (leaflet perforation, etc.)
* Significant tethering of leaflets
* Inflammatory valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who meet the indications and are not contraindicated for treatment by the NeoChord Artificial Chordae Delivery System, Model DS1000.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-02-09 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Level of Mitral Regurgitation Following the Index Procedure | Completion of Index Procedure
  Level of mitral regurgitation per echocardiography

SECONDARY OUTCOMES:
Level of Mitral Regurgitation at 3-6 Months | 3-6 Months
  Level of mitral regurgitation per echocardiography
Level of Mitral Regurgitation at 1 Year | 1 Year
  Level of mitral regurgitation per echocardiography
Level of Mitral Regurgitation at 2 Years | 2 Years
  Level of mitral regurgitation per echocardiography
Level of Mitral Regurgitation at 3 Years | 3 Years
  Level of mitral regurgitation per echocardiography
Level of Mitral Regurgitation at 4 Years | 4 Years
  Level of mitral regurgitation per echocardiography
Level of Mitral Regurgitation at 5 Years | 5 Years
  Level of mitral regurgitation per echocardiography

OTHER OUTCOMES:
Freedom from Mitral Valve Re-intervention | From enrollment until date of mitral valve reintervention, up to 5 years
Freedom from All-Cause Mortality | From enrollment until date of death, up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andres Beiras Fernandez, MD PhD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (5):
- Germany (3):
  - University of Bonn, Bonn
  - CVC Frankfurt, Frankfurt
  - University of Mainz, Mainz
- Hippokration Hospital, Athens, Greece
- Triemli Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No